## MC1481 / 15-004991

Minimal Residual Disease Eradication With Ibrutinib Therapy (MERIT) in Patients With Chronic Lymphocytic Leukemia After Frontline Therapy

NCT02649387

Document Date: 03/12/2021



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

# RESEARCH PARTICIPANT CONSENT AND PRIVACY AUTHORIZATION FORM

**Study Title:** MC1481: Minimal residual disease Eradication with Ibrutinib Therapy (MERIT)

in patients with chronic lymphocytic leukemia after frontline therapy

**IRB#:** 15-004991

Principal Investigator: Asher Chanan-Khan, M.D. and Colleagues

Please read this information carefully. It tells you important things about this research study. A member of our research team will talk to you about taking part in this research study. If you have questions at any time, please ask us.

Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you make your decision.

To help you decide if you want to take part in this study, you should know:

- Taking part in this study is completely voluntary.
- You can choose not to participate.
- You are free to change your mind at any time if you choose to participate.
- Your decision won't cause any penalties or loss of benefits to which you're otherwise entitled.
- Your decision won't change the access to medical care you get at Mayo Clinic now or in the future if you choose not to participate or discontinue your participation.

For purposes of this form, Mayo Clinic refers to Mayo Clinic in Arizona, Florida and Rochester, Minnesota; Mayo Clinic Health System; and all owned and affiliated clinics, hospitals, and entities.

If you decide to take part in this research study, you will sign this consent form to show that you want to take part. We will give you a copy of this form to keep. A copy of this form will be put in your medical record.

IRB#: 15-004991 00 eSign  IRB Doc. Ctrl # 10013.26



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## **CONTACT INFORMATION**

| You can contact | At | If you have questions about |
|---|---|---|
| Principal Investigator: Asher Chanan-Khan, M.D. | <b>Phone:</b> (904) 953-7290 | <ul> <li>Study tests and procedures</li> <li>Research-related injuries or emergencies</li> </ul> |
| | Address:<br>Mayo Clinic Florida | <ul> <li>Any research-related concerns or complaints</li> </ul> |
| | 4500 San Pablo Rd<br>Jacksonville, FL 32224 | <ul><li>Withdrawing from the research study</li><li>Materials you receive</li></ul> |
| | <b>Phone:</b> (904) 308-7300 | <ul> <li>Research-related appointments</li> </ul> |
| | Address: | |
| | St. Vincent's Healthcare 1 Shircliff Way Jacksonville, FL 32204 | |
| Mayo Clinic<br>Institutional Review<br>Board (IRB) | Phone:<br>(507) 266-4000<br>Toll-Free:<br>(866) 273-4681 | Rights of a research participant |
| Research Subject | Phone:<br>(507) 266-9372<br>Toll-Free: | <ul> <li>Rights of a research participant</li> <li>Any research-related concerns or complaints</li> </ul> |
| Advocate<br>(The RSA is independent<br>of the Study Team) | (866) 273-4681<br><b>E-mail:</b> | <ul> <li>Use of your Protected Health<br/>Information</li> </ul> |
| | researchsubjectadvocate@mayo.edu | <ul> <li>Stopping your authorization to use your<br/>Protected Health Information</li> </ul> |
| <b>Patient Account Services</b> | <b>Toll-Free:</b> (844) 217-9591 | Billing or insurance related to this research study |

#### **Other Information:**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## 1. Why are you being asked to take part in this research study?

You are being asked to take part in this research study because you have a lymphoproliferative malignant disorder that remains incurable in the majority of the patients when using standard therapeutic approaches.

The plan is to have about 35 people take part in this study at Mayo Clinic.

## 2. Why is this research study being done?

This research is being done to assess the eradication of minimal residual disease or MRD as well as the toxicity associated with Ibrutinib used as maintenance therapy in Chronic Lymphocytic Leukemia (CLL) patients who achieve a partial response (PR) or complete response (CR) post-induction therapy but who have residual disease (i.e. MRD positive).

The design of this clinical trial allows enrollment of all patients who have completed their initial induction regimen independent of the type of regimen (therapy) given to them as long as they are MRD<sup>+</sup>. Thus, this study will be able to determine prospectively if attainment of MRD<sup>-</sup> post-induction can potentially be possible with the novel agent Ibrutinib given in a *primary* maintenance setting. Thus, this study is unique in following manner (a) it will evaluate the role of single agent Ibrutinib in eradication of MRD; (b) it will evaluate whether the attainment of MRD negativity is possible with Ibrutinib and is it independent of the frontline therapy given; (c) the role and benefit of continuous therapy independent of attainment of MRD negativity and the impact of this in durability of MRD<sup>-</sup> status.

## 3. Information you should know

#### Who is Funding the Study?

Pharmacyclics LLC is funding the study. Pharmacyclics LLC will pay the institution to cover costs related to running the study.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## 4. How long will you be in this research study?

You will continue to receive treatment on this study for up to 3 years, until your disease gets worse, you experience a bad side effect, or you decide not to continue treatment. You will be followed for up to 5 years from the time you start this study so that the researchers can watch your health status.

## 5. What will happen to you while you are in this research study?

If you are eligible to be in the study, you will take Ibrutinib by mouth on days 1-28 of each cycle. Each cycle is 4 weeks. A maximum of 36 cycles of maintenance cycles will be given as long as your disease continues to benefit from the drug and you are not experiencing any bad side effects.

You will be given a diary to record when you take your oral study drug. You will be asked to return your diary, empty pill bottle or any remaining capsules at the end of each cycle.

Before you start treatment, you will begin by completing screening tests that will help to determine if you are able to participate in the study. These tests will include:

- Routine physical exams
- Routine blood tests
- CT scan to document tumor size as a standard assessment for your disease
- EKG and/or ECHO to check the health of your heart. This will only be required if necessary for the routine care of your health
- Routine Bone marrow biopsy and/or aspirate to assess if you have disease present in the bone marrow and to accurately categorize response of your disease prior to treatment given.
- Pregnancy test (only for women able to have children). This will be done within 7 days of starting study drug
- Research blood sample
- Research bone marrow aspirate collection this will only be done if you are scheduled to have your routine bone marrow biopsy.
- DNA sample which may be obtained from one of the following sources: buccal swab (brush the inside of your cheek to collect DNA cells), a skin biopsy (also called a punch biopsy), or myeloid cells from a recent bone marrow



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

If you are found to be a good candidate for the study, you will be expected to complete the following on day 1 of every cycle:

- Routine physical exam (Cycle 7 and onward, you will only be required to come in for physical exams every 3 cycles. You may be seen more often if clinically necessary).
- Adverse event assessment
- Routine blood tests
- Research blood sample

3-4 weeks after your last cycle of treatment you will be expected to complete the following:

- Routine physical exam
- Adverse event assessment
- Routine blood tests
- Bone marrow biopsy and/or aspirate. This will only be done as part of routine care for your disease to evaluate if you have reached complete remission and will be decided by your treating physician
- CT scans
- Research blood sample
- Research bone marrow aspirate. A separate sample will only be collected if you were to have a routine bone marrow biopsy to determine if you have achieved complete remission. A special extra aspirate of the bone marrow will only be required if your blood does not show any evidence of leukemia and to confirm that your bone marrow has also gone into remission. This test is call MRD (or minimal residual disease) assessment and is done to confirm that all detectable disease is cleared

After completing treatment, you will be expected to complete the following every 3 months for 2 years:

- Routine physical exam
- Adverse event assessment
- Routine blood tests
- Bone marrow biopsy and/or aspirate. This will only be done as part of routine care for your disease to evaluate if you have reached complete remission and will be decided by your treating physician
- Research blood sample
- Research bone marrow aspirate.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## 6. What are the possible risks or discomforts from being in this research study?

Many side effects go away shortly after the Ibrutinib is stopped, but in some cases side effects can be serious, long lasting, or may never go away. There may be a risk of death. Some side effects may not be known. Side effects may range from mild to life-threatening. Other drugs may be given to make side effects less serious and less uncomfortable. Talk to the researcher and/or your healthcare provider about side effects and ask any other questions.

#### **Ibrutinib**

**Likely Risks of Ibrutinib** (events occurring in at least 1 of every 5 patients, equal to or more than 20% of the time)

- Occurrence or increase in frequency of loose or watery stools (Diarrhea)
- Muscle and bone pain (Musculoskeletal pain)
- Low white blood cell count (cells that help fight infection) (Neutropenia)
- Rash
- Low platelet count (cells that help blood to clot) (Thrombocytopenia)
- Bleeding (Haemorrhage)
- Nausea
- Fevers

**Less likely risks of Ibrutinib** (events occurring in at least 1 of every 10 patients, equal to or more than 10% of the time)

- Throwing up (Vomiting)
- Headache
- Difficulty passing stool (Constipation)
- Muscle and joint pains (arthralgias)
- Muscle spasms
- Swelling of the hands and feet (Peripheral edema)
- Sensation of lightheadedness or vertigo (spinning sensation) (Dizziness)
- Infection of the lungs (Pneumonia)
- Increase in blood pressure (Hypertension)
- Sores in the mouth
- Common cold (Upper respiratory tract infection)
- Urinary tract infection



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

- Skin infection
- Weakness, tingling, numbness, and pain from nerve damage, usually in the hands and feet (Peripheral neuropathy)

Rare but serious risks of Ibrutinib (events occurring in at least 1 of every 100 patients, equal to or more than 1% of the time)

- Sinus infection (Sinusitis)
- Increase level of "creatinine" in the blood (blood creatinine increased)
- An irregular heartbeat that results from the top/upper chambers of the heart "quivering" instead of beating normally (Atrial fibrillation)
- Blurry vision
- Increased level of uric acid in the blood
- Non-melanoma skin cancer
- Dry mouth
- Increase in specific white blood cell counts (Leukocytosis, Lymphocytosis)
- Low white blood cell counts with fever (febrile neutropenia)
- Skin redness
- Breaking of nails
- Inflammation within the lungs that may lead to permanent damage (Interstitial lung disease)
- Severe infection throughout the body

Heart failure (cardiac failure)

## Side effects that have been seen in less than 1 of every 100 (<1%) patients include:

- Rapid breakdown of cancer cells which releases chemicals and may lead to reduced kidney function. Accumulation of these chemicals may harm muscle or nerve function (Tumor lysis syndrome)
- Itchy rash (Urticaria)
- Inflammation of the fatty tissue underneath the skin (panniculitis)
- Swollen face, lip, mouth, tongue, or throat (Angioedema)
- High WBC count with abnormal clumping that can lead to bleeding (Leukostasis syndrome)
- Severe rash with blisters and peeling skin, particularly around the mouth, nose, eyes, and genitals (Stevens-Johnson syndrome)
- Liver deterioration or failure
- Abnormal rapid and/or irregular heart rhythm that starts from the lower chambers (ventricles) of the heart (Ventricular tachyarrhythmia)
- Temporary or permanent decrease of brain or nerve function due to reduced blood flow to the brain (mini-stroke or stroke)



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

• Tender or painful bumps or ulcers on the skin, sometimes with a fever (Neutrophilic dermatosis)

#### Other Possible risks

Most of these side effects listed above have been mild to moderate in severity; however severe side effects have occurred. Some side effects have been severe enough to lead to study drug discontinuation, dose modification or reduction, hospitalization, disability, and sometimes death.

You should tell your study doctor or medical team about any side effects you are having. Your study doctor may be able to give you medications to help treat the side effects and prevent them from becoming worse. Your study doctor may also choose to stop Ibrutinib for a short time or reduce its dose to allow you to recover from any side effects.

#### Bleeding

You may experience bruising or nosebleeds during treatment with Ibrutinib. Rarely, serious internal bleeding, such as bleeding in your stomach, intestine, or brain may occur, sometimes resulting in death. If you take other medicines or supplements that increase your risk of bleeding, such as aspirin, non-steroidal anti-inflammatory drugs (NSAIDs) or medicines used to prevent or treat blood clots or stroke, Ibrutinib may increase this risk. Blood thinners such as warfarin or other vitamin K antagonists should not be taken together with Ibrutinib. Supplements such as fish oil and vitamin E preparations should be avoided while taking Ibrutinib. Call your study doctor if you have signs or symptoms of serious bleeding, such as blood in your stools or urine or bleeding that lasts for a long time or that you cannot control.

#### Effects on the heart

Abnormal heartbeats and/or irregular heart rhythm (atrial fibrillation, atrial flutter, and/or ventricular tachyarrhythmia) and heart failure, including some fatal events, have been reported in patients treated with Ibrutinib, especially when they also have heart conditions, increased blood pressure, infections, or had abnormal heartbeat in the past You should tell your study doctor immediately if you have any symptoms of heart problems such as feeling as if your heartbeat is fast and irregular, lightheadedness, dizziness, shortness of breath, chest discomfort, swollen legs, or you faint.

#### Infections

You may experience viral, bacterial, or fungal infections during treatment with Ibrutinib. Some of these infections have led to hospitalization and death. Contact your study doctor if you have fever, chills, weakness, confusion, body aches, cold or flu symptoms, vomiting, jaundice, feel tired or feel short of breath - these could be signs of an infection. Your study doctor may start or continue medication to help prevent or treat an infection.

IRB#: 15-004991 00 eSign  IRB Doc. Ctrl # 10013.26



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

A rare and usually fatal viral disease in the brain, Progressive Multifocal Leukoencephalopathy (PML), has been reported in patients treated with Ibrutinib in combination with rituximab and in patients who were previously treated with rituximab. If you experience symptoms such as weakness, paralysis, vision loss and/or impaired speech, you should tell your study doctor immediately.

#### Lymphocytosis and leukostasis

You may experience an increase in the number of lymphocytes, a specific type of white blood cell, in your blood (lymphocytosis). This may occur in the first few weeks of treatment and you should not assume that this increase in white blood cells means that your disease is worsening. This increase may last for several weeks to months. In rare cases, increased number of white blood cells in your bloodstream may alter blood flow resulting in bleeding or clotting (leukostasis). Isolated cases of these events have been reported in patients treated with Ibrutinib. Your study doctor will monitor your blood counts and may administer additional therapy as needed. Talk to your study doctor about what your test results mean.

#### Decreased blood counts

Severe decreases in white blood cells, red blood cells, and platelets (neutropenia, anemia, and thrombocytopenia) were reported in subjects treated with Ibrutinib. If you experience symptoms such as fever, weakness, or easy bruising and/or bleeding, you should tell your study doctor immediately.

#### Allergic reactions

Sometimes people have allergic reactions to drugs. Serious allergic reactions can be life-threatening. If you have an allergic reaction to Ibrutinib, you might develop a rash, difficulty breathing, wheezing when you breathe, sudden low blood pressure with light-headedness, swelling around the mouth, throat or eyes, a racing heartbeat, and/or sweating.

Before starting the study drug, you must tell your study doctor about any drug allergies. You should tell the study doctor right away if you have any allergy symptoms listed above.

#### Rash

A maculopapular rash (flat, red areas on the skin with small bumps) has been commonly reported in patients treated with Ibrutinib alone or in combination with other drugs. Most rashes are mild to moderate in severity and begin 2 to 3 weeks or longer after starting Ibrutinib.

There have been rare reports of severe skin reactions (involving more than 50% of the body) or rash with blisters and peeling skin, which may include open ulcers or sores in the mouth and other areas (Stevens - Johnson syndrome). This could be life-threatening. You should notify your study doctor immediately if you develop a rash that spreads quickly, or if you notice peeling of your skin, with or without ulcers or sores in your mouth.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

#### Non-Melanoma Skin Cancer and Other Cancers

Non-melanoma skin cancer (basal cell carcinoma and squamous cell carcinoma of the skin) have been reported with more frequency and may be related to the use of ibrutinib. Other cancers have been reported such as solid tumors and blood cancers, the relationship to the use of ibrutinib is unknown. You should tell your study doctor if you develop a new cancer while in the study.

#### <u>Tumor Lysis Syndrome (TLS)</u>

Unusual levels of chemicals in the blood caused by the fast breakdown of cancer cells have happened during treatment of cancer and sometimes even without treatment. This may lead to changes in kidney function, abnormal heartbeat, or seizures. Your study doctor may do blood tests to check for TLS.

#### Hypertension

Hypertension is also called high blood pressure and has been commonly reported in subjects treated with ibrutinib. Sometimes, people with high blood pressure may have headaches, dizziness, nervousness, sweating, difficulty in sleeping, facial flushing, or nosebleeds, but in some cases, there may be no symptoms and it may go undetected. After starting ibrutinib, your doctor may measure your blood pressure regularly. You should let your study doctor know if you have any of the symptoms of high blood pressure which may mean that you have developed hypertension or that your hypertension is getting worse. Your study doctor may adjust existing anti-hypertensive medications and/or initiate anti-hypertensive treatment as appropriate.

#### Stroke

Cases of stroke, with and without changes in heartbeat rhythm and/or hypertension have been reported with the use of ibrutinib. Some of these cases have led to death. Seek immediate medical attention if you notice or someone notices in you: sudden numbness or weakness in the limbs (especially on one side of the body), sudden confusion, trouble speaking or understanding speech, sight loss, difficulty walking, loss of balance or lack of coordination, sudden severe headache with no known cause. These may be signs and symptoms of stroke.

#### Liver Failure

Rare cases of liver failure have been reported in patients treated with Ibrutinib. Symptoms of liver failure include yellowing of the eyes and skin (jaundice), itching of the skin, dark colored urine, gray or clay-colored stools, confusion, nausea, loss of appetite, and fatigue or diarrhea. You should tell your study doctor immediately if you have any of these symptoms which may suggest liver disease. Your study doctor may be able to diagnose and provide you required medical care.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

#### Interference with other drugs

Some foods like grapefruit juice and Seville oranges, as well as some medications, may interfere with the way your body processes Ibrutinib. This interference could cause the amount of Ibrutinib in your body to be higher or lower than expected. It is also possible that taking the study drug with your regular medications or supplements, including fish oil, Vitamin E, or other vitamins, may change how your regular medications, or your regular supplements, work. It is very important that you avoid grapefruit juice and Seville oranges and tell the study doctor about all medications, supplements, or herbal medicine like St. John's wort that you are taking during the study. You should notify your study doctor immediately about any side effects to avoid possible harm.

## Drug interruption for any surgical procedures

Ibrutinib may increase the risk of bleeding with any surgical procedure. Ibrutinib should be held at least 3 to 7 days before and after surgery depending upon the type of surgery and the risk of bleeding. Please contact your study doctor if you have any planned surgical procedures. For emergency surgical procedures, Ibrutinib should be discontinued (stopped) after the procedure until the surgical site is reasonably healed (not oozing fluid).

Please contact your study doctor as soon as possible and your study doctor will tell you when to stop Ibrutinib and when to restart it following a surgical procedure.

In addition to the risks listed above, there could be unknown or unexpected side effects associated with the use of Ibrutinib. You will be told in a timely manner, verbally and in writing, of any new information, findings, or changes to the way the research will be done that might influence your willingness to continue your participation in this study.

You may have all, some, or none of the listed side effects of Ibrutinib. Your study doctors and nurses will check you closely for side effects. You may receive medicines or other treatments to prevent or reduce some of these effects. Please tell the study doctor or study staff right away if you have any side effects. Please tell them if you have any other problems with your health or the way you feel during the study, whether or not you think they are related to the study drug.

You should get medical help and contact the study doctor or study staff if you have any of these or any other side effects during the study.

#### Reproductive effects

The effects of Ibrutinib on a developing baby are unknown; therefore women who are pregnant or nursing are not allowed to be in this study. Nobody knows what these risks are right now. Some drugs cause women to have their babies prematurely (early) or to have babies with birth defects.

IRB#: 15-004991 00 eSign  IRB Doc. Ctrl # 10013.26



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

If you are able to have children, you must use a highly effective method of birth control and a barrier method, sexual abstinence, while taking study treatment, as well as for 1 month (women) or 3 months (men) after you stop taking study treatment, to prevent pregnancy in either you or your partner. A "highly effective method of birth control" is defined as a method that has a low failure rate (i.e., less than 1% per year) when used consistently and correctly and includes implants, injectables, birth control pills with 2 hormones, some intrauterine devices (IUDs), sexual abstinence (which is defined as refraining from all aspects of sexual activity) or a sterilized partner. If you are using hormonal contraceptives such as birth control pills or devices, a second barrier method of contraception (e.g., condoms) must be used.

Note: Some birth control pills may not work when you are taking certain drugs. If you have any questions about this, please discuss this with the study doctor.

Be aware that you can still become pregnant even if you use a highly effective method of birth control.

Men: If your partner becomes pregnant while you are on study treatment, or within 3 months of your last dose of Ibrutinib, you must notify the study staff. The study staff will discuss this with you further. You should not donate sperm while you are taking the study drug and for 3 months after you stop taking the study drug.

Women: If you become pregnant while you are on study treatment or within 1 month of your last dose of Ibrutinib you must notify the study staff. If you become pregnant on the study, you must immediately stop taking the study treatment. The Sponsor will continue to collect information about your pregnancy and the birth of your baby even after study treatment is stopped.

## Breast-feeding

It is not known whether ibrutinib or its metabolites are excreted in human milk. Because many drugs are excreted in human milk and because of the potential for serious adverse reactions in nursing infants from ibrutinib, breast-feeding should be discontinued during ibrutinib treatment.

## 7. Are there reasons you might leave this research study early?

You may decide to stop at any time. You should tell the Principal Investigator if you decide to stop and you will be advised whether any additional tests may need to be done for your safety.

In addition, the Principal Investigator or Mayo Clinic may stop you from taking part in this study at any time:

• if it is in your best interest,



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

- if you don't follow the study procedures,
- if you are not benefiting from the study treatment,
- if the study is stopped.

If you leave this research study early, or are withdrawn from the study, no more information about you will be collected; however, information already collected about you in the study may continue to be used.

We will tell you about any new information that may affect your willingness to stay in the research study.

## 8. What if you are injured from your participation in this research study?

#### Where to get help:

If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the beginning of this form. Mayo Clinic will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

#### Who will pay for the treatment of research related injuries?

Care for such research-related injuries will be billed in the ordinary manner, to you or your insurance. You will be responsible for all treatment costs not covered by your insurance, including deductibles, co-payments and coinsurance.

## 9. What are the possible benefits from being in this research study?

Over 25 clinical trial evaluations have been completed and established the importance of minimal residual disease (MRD). Analyses of these clinical studies have demonstrated a significant progression free survival (PFS) benefit among patients who have achieved MRD-negative (MRD) state. Patients who are in CR and are MRD tend to have up to 2 years advantage in PFS vs. those who are in CR and maintain residual detectable disease. Collectively, the data suggests that attainment of MRD disease after first-line therapy may have an important impact on the clinical outcome of patients with CLL.

IRB#: 15-004991 00 eSign  IRB Doc. Ctrl # 10013.26



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## 10. What alternative do you have if you choose not to participate in this research study?

You do not have to be in this study to receive treatment for your Chronic Lymphocytic Leukemia. Your other choices may include:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting no treatment
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

You should talk to the researcher and your regular physician about each of your choices before you decide if you will take part in this study.

## 11. What tests or procedures will you need to pay for if you take part in this research study?

You won't need to pay for tests and procedures which are done just for this research study. These tests and procedures are:

- Study drug, Ibrutinib
- Research tests done on your blood, saliva, bone marrow and skin biopsy

However, you and/or your insurance will need to pay for all other tests and procedures that you would have as part of your clinical care. These tests and procedures are:

- Routine exams and blood tests
- Routine bone marrow biopsy and aspirate for your disease assessment
- CT scans
- EKG/ECHO
- Pregnancy test for women of childbearing potential

You will also be responsible for any co-payments and deductibles.

If you have billing or insurance questions call Patient Account Services at the telephone number provided in the Contact Information section of this form.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

## 12. Will you be paid for taking part in this research study?

You will not be paid for taking part in this study. You will not receive any compensation for or benefit from any patents or discoveries that may result from your participation in this research study.

## 13. What will happen to your samples?

We would like to keep your research samples for future research. You can still take part in this current study even if you don't want your sample used for future research. If you agree to give your sample, it will be the property of Mayo Clinic.

Other researchers at Mayo Clinic who aren't involved with this study may ask to use your sample for future research. Researchers at other institutions may also ask for a part of your sample for future studies. Your sample will be sent to researchers in a coded format, which protects your identity.

Some future studies may examine your DNA, which is the genetic information you inherited from your parents (genetic testing). The Principal Investigator may contact you if there are findings which may be useful for your health care. You would be given general information on the potential risks, benefits, and costs of choosing to learn about the findings.

## Please read the following statements and mark your choices:

| 1. | I permit my sample to be stored and used in future research of CLL at Mayo Clinic: | | |
|---|---|---|---|
| | Yes | ☐ No | Please initial here: |
| 2. | . I permit my sample to be stored and used in future research at Mayo Clinic to learn abou prevent, or treat any other health problems: | | |
| | Yes | ☐ No | Please initial here: |
| 3. | . I permit Mayo Clinic to give my sample to researchers at other institutions: | | |
| | Yes | ☐ No | Please initial here: |



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

There is a very small chance that some commercial value may result from the use of your donated sample. If that happens, you won't be offered a share in any profits.

You may request to have your sample destroyed by writing to the Principal Investigator. The address is found in the "Contact Information" section of this consent form.

Because we cannot predict how your sample will be used in the future, we cannot promise that samples can be retrieved and destroyed.

## 14. How will your privacy and the confidentiality of your records be protected?

Mayo Clinic is committed to protecting the confidentiality of information obtained about you in connection with this research study.

By signing this form, you authorize Mayo Clinic and the investigators to use and disclose any information created or collected in the course of your participation in this research protocol. This information might be in different places, including your original medical record, but we will only disclose information that is related to this research protocol for the purposes listed below.

To protect the data and confidentiality of subjects' data, a code will be used as an identifier. The code will be a registration number assigned specifically to the patient by the Mayo Clinic Cancer Center Registration Office or Study Sponsor, if applicable. The correlating Mayo Clinic number and the patient's name for reference will be maintained in a secure database accessible by Mayo Clinic assigned research staff. All information will be de-identified removing names and any clinical data markers that are linked to the patient. Study files will be maintained in the secure research area and only staff assigned to this project will have access to those files. Data and samples will be coded with numbers, study-related research materials will be locked in cabinets, and data will be password-protected stored on a computer. The patient's confidentially will be protected by complying with all Mayo Clinic and IRB rules. The principal investigator will carefully monitor the study for any developing risks or adverse events and report them immediately to the IRB. Any records needed by monitor will be copied by coordinator to ensure that all identifying information is redacted. If the results of the research are made public, information that identifies you will not be used.

Representatives from the Mayo Clinic Institutional Review Board (the committee that reviews, approves, and monitors research on human subjects) may inspect study records during internal auditing procedures. However, these individuals are required to keep all information confidential.

IRB#: 15-004991 00 eSign  IRB Doc. Ctrl # 10013.26



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

During this research, information about your health will be collected. Under Federal law called the Privacy Rule, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use and share your health information for research and why they may need to do so. Information about you and your health cannot be used in this research study without your written permission. If you sign this form, it will provide that permission.

#### Health information may be collected about you from:

- Past, present and future medical records.
- Research procedures, including research office visits, tests, interviews and questionnaires.

### Why will this information be used and/or given to others?

- To do the research.
- To report the results.
- To see if the research was done correctly.

If the results of this study are made public, information that identifies you will not be used.

## Who may use or share your health information?

- Mayo Clinic research staff involved in this study.
- Pharmacyclics LLC, its affiliates, and its collaborators (e.g. Janssen Biotech, Inc.)

#### With whom may your health information be shared?

- The Mayo Clinic Institutional Review Board that oversees the research.
- Other Mayo Clinic physicians involved in your clinical care.
- Researchers involved in this study at other institutions.
- Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health, and other United States agencies) or government agencies in other countries that oversee or review research.
- The sponsor(s) of this study and the people or groups it hires to help perform this research.
- A group that oversees the data (study information) and safety of this research.

In addition, individuals involved in study oversight and <u>not</u> employed by Mayo Clinic may be allowed to review your health information included in past, present, and future medical and/or research records. This review may be done on-site at Mayo Clinic or remotely (from an off-site location). These records contain information that directly identifies you. However, the individuals will not be allowed to record, print, or copy (using paper, digital, photographic, or other methods), or remove your identifying information from Mayo Clinic.



Approval Date: March 12, 2021 Not to be used after: January 26, 2022

#### Is your health information protected after it has been shared with others?

Mayo Clinic asks anyone who receives your health information from us to protect your privacy; however, once your information is shared outside Mayo Clinic, we cannot promise that it will remain private and it may no longer be protected by the Privacy Rule.

## **Your Privacy Rights**

You do not have to sign this form, but if you do not, you cannot take part in this research study.

If you cancel your permission to use or share your health information, your participation in this study will end and no more information about you will be collected; however, information already collected about you in the study may continue to be used.

If you choose not to take part or if you withdraw from this study, it will not harm your relationship with your own doctors or with Mayo Clinic.

You can cancel your permission to use or share your health information at any time by sending a letter to the address below:

Mayo Clinic
Office for Human Research Protection
ATTN: Notice of Revocation of Authorization
200 1st Street SW
Rochester, MN 55905

Alternatively, you may cancel your permission by emailing the Mayo Clinic Research Subject Advocate at: researchsubjectadvocate@mayo.edu.

Please be sure to include in your letter or email:

- The name of the Principal Investigator,
- The study IRB number and /or study name, and
- Your contact information.

Your permission lasts forever, unless you cancel it.



Signature

Name and Clinic Number

Approval Date: March 12, 2021 Not to be used after: January 26, 2022

| ENROLLMENT AND PERMISSION SIGNATURES Your signature documents your permission to take part in this research. | | |
|---|---|---|
| Signature | | |
| - | ent<br>ne research study to the participant.<br>Il questions about this research study to t | the best of my ability. |
| Printed Name | Date (mm/dd/yyyy) | Time (hh:mm am/pm) |